CLINICAL TRIAL: NCT06494826
Title: Decoding the Clinical Impact of Host and Microbial Intestinal Proteomic Landscape in Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Weizmann Institute of Science (Other)
Collaborators: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0078-23-EMC
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool samples blood samples gastrointestinal brushes gastrointestinal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- crohn disease patients: Candidates for a medically-indicated, diagnostic colonoscopy due to suspected new-onset CD.
  Interventions: Other: colonoscopy procedure
- healthy controls: healthy participants admitted for non-specific GI complaints (such as changes in bowel movements, bloating, abdominal pain) or routine screening for colorectal cancer as part of primary
  Interventions: Other: colonoscopy procedure

INTERVENTIONS:
Other: colonoscopy procedure — Candidates for a medically-indicated colonoscopy due to suspected new-onset CD or non-specific GI complaints or routine screening for colorectal cancer as part of primary prevention.
  colonoscopy will not be done for research purposes only .

SUMMARY:
In this study, the investigators will explore our protein-based platform assessing commensals potentially contributing to features of CD, while assessing the global composition and abundance of AMPs expressed in the GI tract under specific CD-relevant clinical contexts. This would enable us to (a) identify new commensals contributing to features of CD spectrum and various sub-types; (b) uncover the mechanistic basis of dysbiosis in CD (c) utilize the pipeline to develop new theranostic for disease exacerbation, complication and treatment responses; and (d) potentially enable future exploitation of novel AMP combinations, and their respective antimicrobial capacity to counteract dysbiosis in CD.

Uncovering the proteomic manifestations of perturbed host-microbiome communications in CD will eventually enable the development and validation of clinical non-invasive surrogate markers, mechanistically determine causative drivers of CD, and potentially facilitate the development of novel therapeutic interventions.

DETAILED DESCRIPTION:
Participants will be recruited from a community outpatient clinics and from a leading outpatient gastroenterology clinic: Emek Medical Center, after ICF signing , they will fill out a medical, demographic, and lifestyle habits questionnaires, as well as a food frequency questionnaire (FFQ). Participants will receive a home stool kit and will be instructed on how to use it. They will also receive a kit and an explanation regarding preparation materials for the colonoscopy. Subjects will be asked to collect stool samples at home - prior to colonoscopy and if possible - after colonoscopy bowel prep.

The seconed visit of the study will occure on the day of colonoscopy. Each patient will be clinically assessed by a gastroenterologist using the Crohn's Disease Activity Index (CDAI)30 and Harvey-Bradshaw Index (HBI); and collection of luminal, brush cytology, and mucosal samples from 4 different lower intestine regions

ELIGIBILITY:
Inclusion criteria - CD study group:

* Age ≥ 18
* Candidates for a medically-indicated, diagnostic colonoscopy due to suspected new-onset CD.
* Naïve to any medical or nutritional intervention.

Inclusion criteria - healthy controls:

• Age- and gender-matched patients to the CD group, admitted for non-specific GI complaints (such as changes in bowel movements, bloating, abdominal pain) or routine screening for colorectal cancer as part of primary prevention per clinical guidelines.

Exclusion Criteria - both groups:

* Established diagnosis of inflammatory bowel disease (IBD) with prior treatment.
* Chronic gastro-intestinal disorder (e.g. celiac disease, eosinophilic esophagitis, collagenous gastritis, autoimmune gastritis, etc.).
* Type 1 or type 2 diabetes mellitus.
* Past or present history of malignancy.
* BMI > 30 (kg/m2)
* Use of systemic antibiotics or probiotics 2 months prior to enrolment.
* Use of steroids 2 months prior to enrolment (not including a short course of topical steroidal therapy).
* Any previous major gastric or intestinal surgery.
* Suspected or proven extensive involvement of non-ileal small intestine or colon, or significant perianal disease.
* Significantly stricturing or penetrating (fistulizing) disease at presentation.
* Chronic treatment with any oral/systemic immunosuppressive or anti-inflammatory drugs (e.g. steroids, 5-aminosalicylic acid, immunomodulators, biologics, etc.). Patients receiving these drugs as inhalers/creams/ointments should not be excluded from the study.
* Primary immunodeficiency.
* Pregnancy or breastfeeding in the last 6 months.
* Serious medical conditions that may alter the gut microbiome composition, based on investigators judgement (for example primary immunodeficiency, autoimmune disorder, or rheumatologic disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CD study group will consist of candidates for a medically-indicated, diagnostic colonoscopy due to suspected new-onset CD.
  Naïve to any medical or nutritional intervention. for healthy controls: Age- and gender-matched patients to the CD group, admitted for non-specific GI complaints (such as changes in bowel movements, bloating, abdominal pain) or routine screening for colorectal cancer as part of primary prevention per clinical guidelines.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Characterization of gut microbiota and associated molecules in Crohn's disease and healthy human gastrointestinal tract | 1 week
  Identification of changes in fecal microbiota and associated molecules using multi-dimensional analysis of fecal samples, biopsies and brushes collected during endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Emek medical center, Afula, Israel